CLINICAL TRIAL: NCT01840852
Title: the Effects of Inflammatory Cytokines on Sleep During Acute Diverticulitis
Brief Title: Sleep and Cytokines During Acute Diverticulitis
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Ismail Gögenür, Senior resident and D.Sc., Herlev Hospital
Other Study IDs: CHU-1
Record Dates: First submitted 2013-04-13; First posted 2013-04-26 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Acute Diverticulitis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- acute uncomplicated diverticulitis: CT-verified acute uncomplicated diverticulitis managed by antibiotics

SUMMARY:
The purpose of this study is to investigate sleep disturbances during Acute uncomplicated diverticulitis by polysomnography. The investigators hypothesis is the inflammation causes REM(rapid eye movement)-sleep reduction and this is correlated with plasma cytokine levels.

DETAILED DESCRIPTION:
An increasing number of experimental studies have showed that inflammation can induce disturbances in sleep architecture, mediated by cytokines. Sleep is important both in health and disease processes and can affect recovery, morbidity and mortality.

Studies have been done on sleep disturbances after major and minor GI-surgery but never in relation to none surgical inflammatory diseases, namely acute diverticulitis.

This study will investigate sleep architecture by Polysomnography and inflammation by levels of pro inflammatory cytokines in plasma.

Following methods will be applied

Device: Polysomnograph - Embla Titanium (Natus Medical Incorporated, USA)

Procedure: Plasma cytokines (IL-2, IL-6 and TNF(tumor necrosis factor-alfa)

Procedure: Plasma CRP(C reactive protein) and leukocytes

ELIGIBILITY:
Inclusion Criteria:

* CT-verified diverticulitis patients managed by antibiotic treatment at Herlev Hospital
* Pain and fever occurred less than 72 hours prior to the admission
* ASA (American Society of Anesthesiologists) score I to III

Exclusion Criteria:

* Surgical intervention needed
* Complicated diverticulitis
* Complications in relation to diverticulitis
* Pain and fever occurred more than 72 hours prior to the admission
* In anticoagulant treatment and heart rate control treatment
* Known Autoimmune disease
* Known medically treated sleep-disorder (insomnia, restless legs etc.) and sleep apnea
* Shift-work or jetlag
* Daily use of opioid, psychopharmaca, opioids or anxiolytics (including Hypnotics)
* Known psychiatry conditions in treatment with psychopharmaca
* Daily alcohol intake of more than 5 units or drug abuse
* Missing written consent
* Diabetes Mellitus
* Predicted bad compliance
* Pregnant or breast-feeding
* Urine or fecal incontinence
* Severe kidney disease
* Current cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 16 x Acute uncomplicated diverticulitis (Hansen and stock stage 1) patients aged 18-75 years managed by antibiotic treatment at Herlev Hospital.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
change in Sleep architecture during acute uncomplicated diverticulitis from baseline at the remission (30th day) | 1st, 2nd and 30th nights following the admission
  Sleep architecture measured by Polysomnography (awake, stadium I-IV, REM sleep, sleep latency, awakenings)
change in cytokine levels in plasma during the acute uncomplicated diverticulitis from baseline levels at remission | 1st, 2nd and 30th nights following the admission
  the Blood sample is taken prior to night sleep; Cytokines are measured by commercial ELISA-kits
change in CRP level in plasma during the acute uncomplicated diverticulitis from baseline levels at remission | 1st, 2nd and 30th nights following the admission
  the Blood sample is taken prior to night sleep; CRP is measured by standardized conventional method
change in leucocyte level in plasma during the acute uncomplicated diverticulitis from baseline levels at remission | 1st, 2nd and 30th nights following the admission
  the Blood sample is taken prior to night sleep; Leucocyte is measured by standardized conventional method

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, M.D., Principal Investigator — University of Copenhagen, Herlev Hospital
Locations (1):
- Department D, Herlev Hospital, Herlev, Copenhagen, Denmark